CLINICAL TRIAL: NCT01251172
Title: Phase II Study of RO4929097 to Eradicate Residual Disease in Patients With Multiple Myeloma Post Single Autologous Stem Cell Transplant
Brief Title: RO4929097 After Autologous Stem Cell Transplant in Treating Patients With Multiple Myeloma
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: Lack of Drug Supply
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NCI-2011-02555; NCI-2011-02555 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); CDR0000689644; 011003 (Other: Rutgers Cancer Institute of New Jersey); 8540 (Other: CTEP); P30CA072720 (NIH); U01CA132194 (NIH)
Record Dates: First submitted 2010-11-30; First posted 2010-12-01 (Estimated); Last update posted 2017-09-28 (Actual); Status verified 2017-09

CONDITIONS: DS Stage I Plasma Cell Myeloma; DS Stage II Plasma Cell Myeloma; DS Stage III Plasma Cell Myeloma; Refractory Plasma Cell Myeloma
MeSH Terms: conditions — Multiple Myeloma | interventions — 2,2-dimethyl-N-(6-oxo-6,7-dihydro-5H-dibenzo(b,d)azepin-7-yl)-N'-(2,2,3,3,3-pentafluoropropyl)malonamide; Hematopoietic Stem Cell Mobilization; Melphalan

ARMS (1):
- Treatment (RO4929097 after autologous stem cell transplant) (Experimental): STEM CELL TRANSPLANTATION AND CHEMOTHERAPY: Patients undergo standard mobilization and collection of autologous peripheral stem cells (>= 4.0 x 10^6 CD34+ cells/kg). Patients then receive high-dose melphalan IV on days -3 and -2 and undergo autologous stem cell transfusion on day 0. Patients with progressive disease, stable disease, partial response, stringent complete response, or complete response are taken off study; patients with residual/persistent disease (VGPR) continue to therapeutic treatment.
  THERAPEUTIC TREATMENT: Beginning 100-110 days after transplantation, patients receive oral gamma-secretase inhibitor RO4929097 once daily on days 1-3, 8-10, and 15-17. Courses repeat every 21 days in the absence of disease progression or unacceptable toxicity.
  Interventions: Procedure: Autologous Hematopoietic Stem Cell Transplantation; Drug: Gamma-Secretase Inhibitor RO4929097; Procedure: Hematopoietic Stem Cell Mobilization; Procedure: In Vitro-Treated Peripheral Blood Stem Cell Transplantation; Other: Laboratory Biomarker Analysis; Drug: Melphalan

INTERVENTIONS:
Procedure: Autologous Hematopoietic Stem Cell Transplantation — Undergo in vitro treated autologous peripheral blood stem cell transplant
  Other Names: Autologous Stem Cell Transplantation
Drug: Gamma-Secretase Inhibitor RO4929097 — Given orally
  Other Names: RO4929097
Procedure: Hematopoietic Stem Cell Mobilization — Undergo standard mobilization
Procedure: In Vitro-Treated Peripheral Blood Stem Cell Transplantation — Undergo in vitro treated autologous peripheral blood stem cell transplant
  Other Names: in vitro-treated PBPC transplantation; in vitro-treated peripheral blood progenitor cell transplantation
Other: Laboratory Biomarker Analysis — Correlative studies
Drug: Melphalan — Given IV
  Other Names: Alanine Nitrogen Mustard; CB-3025; L-PAM; L-Phenylalanine Mustard; L-Sarcolysin; L-Sarcolysin Phenylalanine mustard; L-Sarcolysine; Melphalanum; Phenylalanine Mustard; Phenylalanine Nitrogen Mustard; Sarcoclorin; Sarkolysin; WR-19813

SUMMARY:
This phase II clinical trial is studying how well gamma-secretase/Notch signalling pathway inhibitor RO4929097 (RO4929097) after autologous stem cell transplant works in treating patients with multiple myeloma. Giving chemotherapy, such as melphalan, before autologous stem cell transplant stops the growth of cancer cells by stopping them from dividing or killing them. Before treatment, stem cells are collected from the patient's blood and stored. After chemotherapy, the stem cells are returned to the patient to replace the blood-forming cells that were destroyed by the chemotherapy. RO4929097 may stop the growth of cancer cells by blocking some of the enzymes needed for cell growth. Giving RO4929097 after autologous stem cell transplant may kill more cancer cells.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To determine the efficacy of RO4929097 in eradicating residual/persistent disease (conversion of VGPR to CR or sCR status) in multiple myeloma patients status post single high-dose melphalan/autologous stem cell rescue with residual/persistent disease post-transplant.

SECONDARY OBJECTIVES:

I. To determine the safety of single agent RO4929097 post-autologous stem cell transplant in multiple myeloma patients.

II. To analyze Notch receptor and ligand protein expression in pre-transplant, pre-treatment with RO4929097, and post-treatment bone marrow biopsy samples.

III. To isolate and identify clonogenic multiple myeloma progenitor cells from bone marrow aspirate and/or peripheral blood at the following time points: pre-transplant, day 100 post-transplant, and post-treatment staging bone marrow biopsy.

IV. To analyze Notch receptor and ligand protein expression on isolated clonogenic progenitor myeloma cells.

V. To characterize the tumor xenograft-initiating potential of clonogenic myeloma cells in adult Casper zebrafish and SCID-hu model and evaluate the drug toxicity and therapeutic potential of RO4929097 with this model.

VI. To analyze anti-angiogenic effects of RO4929097 as measured by reduction in microvessel density and VEGFR-1 expression in pre-treatment and post-treatment bone marrow biopsy samples.

VII. To determine whether measurement of soluble surrogate markers of angiogenesis prior to and following treatment with RO4929097 provide an early marker of disease response to Notch inhibition.

OUTLINE: This is a multicenter study.

STEM CELL TRANSPLANTATION AND CHEMOTHERAPY: Patients undergo standard mobilization and collection of autologous peripheral stem cells (>= 4.0 x 10^6 CD34+ cells/kg). Patients then receive high-dose melphalan IV on days -3 and -2 and undergo autologous stem cell transfusion on day 0. Patients with progressive disease, stable disease, partial response, stringent complete response, or complete response are taken off study; patients with residual/persistent disease (very good partial response [VGPR]*) continue to therapeutic treatment.

NOTE: *Patients who meet the criteria for VGPR but have findings of abnormal bone marrow cytogenetic study demonstrating >= 10% metaphase cells positive for either high-risk chromosomal abnormalities or persistent disease-related chromosomal abnormalities (e.g., chromosome del 13; del17p, t(4;14), t(14;16), t(6;14) or complex cytogenetics) will have a repeat bone marrow biopsy assessment with cytogenetics within 2-3 weeks. If the repeat biopsy findings suggest persistent high-risk cytogenetic findings, then the patient is considered eligible to receive RO4929097 to eradicate residual disease.

THERAPEUTIC TREATMENT: Beginning 100-110 days after transplantation, patients receive oral RO4929097 once daily on days 1-3, 8-10, and 15-17. Courses repeat every 21 days in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients are followed up for at least 4 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Patients must have a diagnosis of multiple myeloma as defined below with staging based on the International Staging System:

  * Multiple myeloma - all three required (Note: these criteria identify stage 1B and stages II and IIIA/B myeloma by Durie/Salmon stage; stage 1A becomes smoldering or indolent myeloma):

    * Monoclonal plasma cells in the bone marrow ≥ 10% and/or presence of a biopsy-proven plasmacytoma
    * Monoclonal protein present in the serum and/or urine (if no monoclonal protein is detected [non-secretory disease], then >= 30% monoclonal bone marrow plasma cells and/or biopsy-proven plasmacytoma is required)
    * Myeloma-related organ dysfunction (1 or more) (a variety of other types of end organ dysfunctions can occasionally occur and lead to a need for therapy; such dysfunction is sufficient to support classification as myeloma if proven to be myeloma related):

      * Calcium elevation in the blood (serum calcium > 10.5 mg/L or upper limit of normal)
      * Renal insufficiency (serum creatinine > 2mg/dL)
      * Anemia (hemoglobin < 10 g/dL or 2 g < normal)
      * Lytic bone lesions or osteoporosis (if a solitary [biopsy-proven] plasmacytoma or osteoporosis alone [without fractures] are the sole defining criteria, then > 30% plasma cells are required in the bone marrow)
* Patients must have measurable disease

  * Patients with non-secretory multiple myeloma will be eligible only if the baseline serum free light chain level is elevated (>= 10 mg/dL)
* For therapeutic treatment with RO4929097, patients must have peripheral blood stem cell collection of >= 4.0 x 10^6 cells/kg (patient's ideal body weight)
* ECOG performance status =< 2, Karnofsky >= 60%
* Estimated life expectancy of at least 12 weeks
* Absolute neutrophil count (ANC) >= 1,500/mcL
* Platelets >= 100,000/mcL
* Hemoglobin >= 9.0 g/dL
* NOTE: Patients should not require chronic supportive growth factor administration or transfusions to meet treatment eligibility criteria (e.g., G-CSF for ANC eligibility)
* Serum creatinine =< 2.0 mg/dL OR a measured creatinine clearance by 24-hour urine collection >= 40 mL/min (a calculated creatinine clearance by Cockcroft-Gault formula is acceptable in lieu of a measured value)
* Total bilirubin within normal institutional limits
* AST (SGOT)/ALT SGPT) =< 2.5 X institutional ULN
* Patients with uncontrolled electrolyte abnormalities including hypocalcemia, hypomagnesemia, hyponatremia, hypophosphatemia, or hypokalemia, defined as less than the lower limit of normal for the institution despite adequate electrolyte supplementation, are excluded from this study
* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use two forms of contraception (i.e., barrier contraception and one other method of contraception) at least 4 weeks prior to study entry, for the duration of study participation, and for at least 12 months post-treatment
* No requirement for routine use of hematopoietic growth factors (including granulocyte colony-stimulating factor, granulocyte-macrophage colony-stimulating factor, or interleukin-11) or platelet transfusions to maintain absolute neutrophil counts or platelet counts above the required thresholds for study entry

  * Use of erythropoietin-stimulating agents and red cell transfusions are also not permitted prior to initiation of RO4929097
* Patient must meet the institutional standard criteria for undergoing high-dose chemotherapy and autologous stem cell transplant
* No serious concomitant systemic disorders (including active infections) that would compromise the safety of the patient or compromise the patient's ability to complete the study, at the discretion of the investigator
* No uncontrolled intercurrent illness including, but not limited to:

  * Ongoing or active infection
  * Symptomatic congestive heart failure
  * Unstable angina pectoris
  * A history of torsades de pointes
  * Cardiac arrhythmia other than chronic, stable atrial fibrillation
  * Psychiatric illness/social situations that would limit compliance with study requirements
* No baseline QTcF > 450 msec (male) or QTcF > 470 msec (female)
* Patients with malabsorption syndrome, disease significantly affecting gastrointestinal function, or resection of the stomach or small bowel are excluded

  * Subjects with ulcerative colitis, inflammatory bowel disease, or a partial or complete small bowel obstruction are also excluded
* No condition (e.g., gastrointestinal tract disease resulting in an inability to take oral medication or a requirement for IV alimentation, prior surgical procedure affecting absorption, or active peptic ulcer disease) that impairs the ability to swallow and retain RO4929097
* Patients who have active hepatitis B or C, or have a history of liver disease, other forms of hepatitis or cirrhosis are ineligible
* HIV-positive patients on combination antiretroviral therapy are ineligible
* No second primary malignancy except most situ carcinoma (e.g., in situ carcinoma of the of the cervix, adequately treated non-melanomatous carcinoma of the skin) or other malignancy treated at least 3 years previously with no evidence of recurrence
* No history of allergic reactions attributed to compounds of similar chemical or biologic composition to RO4929097or other agents used in the study
* There are no limitations on type and amount of prior therapy with the following exception: patients who have had a solid organ transplant are ineligible

  * Acute toxicities of high-dose melphalan therapy must have resolved to the NCI-CTCAE version 4.0 grade 1 or less (with the exception of alopecia)
* Patients taking medications with narrow therapeutic indices that are metabolized by cytochrome P450 (CYP450), including warfarin sodium (Coumadin®) are ineligible
* No concurrent medications that are strong inducers/inhibitors or substrates of CYP3A4
* No concurrent drugs, food, supplements, or over-the-counter medications that may interfere with the metabolism of RO4929097, including ketoconazole and fresh-squeezed grapefruit juice
* Patients may not be receiving any other investigational agents
* Patients may not be receiving antiarrhythmics or other medications known to prolong QTc
* No other investigational or commercial agents or therapies may be administered with the intent to treat the patient's malignancy
* No patients who have had any chemotherapy or radiotherapy post-autologous stem cell transplant prior to entering the therapeutic arm of the study or those who have not recovered from the high-dose melphalan and autologous stem cell transplant
* For therapeutic treatment with RO4929097, the acute toxicities of the high-dose melphalan therapy must have resolved to the NCI-CTCAE version 4.0 Grade 1 or less (with the exception of alopecia)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2010-12; Primary Completion 2012-07 (Actual)

PRIMARY OUTCOMES:
Overall response rate of gamma-secretase/Notch signalling pathway inhibitor RO4929097 in eradicating residual/persistent disease, defined as conversion from VGPR to CR or sCR | Up to 42 days
  A Simon's 2-stage optimal Phase II design will be used to monitor the study.

SECONDARY OUTCOMES:
Clonogenic myeloma progenitor cells | At baseline, at 100 days post-transplant, and at 6 weeks
  Logistic regression models will be used to study the association of clinical response (relapse) and the myeloma stem cell kinetics (present and absent of cell, and/or percentage of cells).
Incidence of adverse events and abnormal laboratory variables as assessed according to the NCI-CTCAE version 4.0 | Up to 30 days
  Adverse events will be reported in frequency tables overall, by intensity, and by relationship.

CONTACTS AND LOCATIONS:
Overall Officials: Mecide Gharibo, Principal Investigator — Rutgers Cancer Institute of New Jersey
Locations (1):
- Moffitt Cancer Center, Tampa, Florida, United States